CLINICAL TRIAL: NCT05666739
Title: NIEHS Repository of Stored Biological Samples for Future Use
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001073; 001073-E
Record Dates: First submitted 2022-12-24; First posted 2022-12-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05-05

CONDITIONS: Normal Physiology
Keywords: Blood; Urine; Assay Development; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy controls: General public population, including females and males, who are over the age of 18, with a mixture of races and ethnicities representative of North Carolina

SUMMARY:
Background:

Laboratory tests that use blood and urine can provide a great deal of information about human health and disease. To develop even better tests and to improve the ways samples are handled for testing researchers need to experiment with samples from healthy people.

Objective:

This natural history study will collect blood and urine from healthy people. The samples will build a repository that will be used for all kinds of research.

Eligibility:

Healthy people aged 18 years or older.

Design:

Participants will have 1 study visit. The visit will last up to 2 hours.

Participants will be screened. They will answer questions about their health history. They will list any medications they take. They will consent to donate samples for research and future use:

Blood: Up to 4.5 tablespoons of blood may be collected from a needle inserted into a vein.

Urine: Participants will be given a sterile container to provide a sample.

Some participants may be asked to provide other types of samples.

Some participants may be asked to provide new samples if their first ones are depleted.

DETAILED DESCRIPTION:
Study Description:

We aim to build a repository utilizing both prospectively and retrospectively collected human biological samples, like blood and urine, to develop and test the following: specific laboratory assays, to develop and maintain freezer and specimen handling quality control, to have blinded quality control specimens for laboratory testing, and to assess exposure variability over time.

Objectives:

Primary Objective: To build a repository for approved investigators to access stored biological samples for the following: developing and testing specific laboratory assays, to maintain freezer and specimen handling quality control, to have blinded quality control specimens for testing labs, and to assess exposure variability over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for prospective biospecimen collection:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Ability to provide informed consent.
3. Male or female, aged >=18
4. Able to travel to the NIEHS CRU for study visits

EXCLUSION CRITERIA:

Exclusion Criteria for prospective biospecimen collection:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Not willing to have samples stored for future use.
2. Any condition that, in the investigator s opinion, places the participant at undue risk for complications associated with required study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The general community sample will be from Durham, Raleigh, Chapel Hill and other nearby cities close to the NIEHS Clinical Research Unit (CRU).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2032-07-19 (Estimated); Study Completion 2032-07-19 (Estimated)

PRIMARY OUTCOMES:
To build a repository for approved investigators to access stored biological samples for the following: developing and testing specific laboratory assays, to maintain freezer and specimen handling quality control, to have blinded quality control... | On-going
  To build a repository for approved investigators to access stored biological samples for the following: developing and testing specific laboratory assays, to maintain freezer and specimen handling quality control, to have blinded quality control specimens for testing labs, and to assess exposure variability over time.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Kirschner, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Most of the participant data will be utilized by investigators in an aggregate way to validate or invalidate their research.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001073-E.html